CLINICAL TRIAL: NCT05929456
Title: Multispectral and Bimodal Fluorescent Guided Surgery (FGS) of High-grade Glioma for Refining Margin Assessment: A Phase 1 Dose Finding Study Using Cetuximab-IRDye800CW Combined With 5-ALA.
Brief Title: Multispectral Bimodal Fluorescence Guided Surgery of High-grade Glioma With Cetuximab-800CW and 5-ALA (5-aminolevulinic Acid)
Acronym: MIRROR
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NC2022-01
Record Dates: First submitted 2023-05-25; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Glioblastoma; High-grade Glioma
Keywords: Fluorescence guided surgery; Glioblastoma; High-grade glioma; 5-ALA
MeSH Terms: conditions — Glioblastoma; Glioma

STUDY DESIGN:
Intervention Model Description: prospective, single center phase I feasibility and dose finding study in a single cohort, i.e patients with glioblastoma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Glioblastoma group (Experimental): This study will consist of 1 group and therefore 1 arm
  Interventions: Drug: Cetuximab-IRDye800

INTERVENTIONS:
Drug: Cetuximab-IRDye800 — patients will receive a single IV injection of Cetuximab-IRDye800CW 2-4 days prior to surgert. The IMP (Investigational medicinal product)/tracer will be used for fluorescence guided surgery.

SUMMARY:
The MIRROR study is a prospective, single center phase I feasibility and dose finding study in patients with high-grade glioma, to establish the safety, feasibility, and optimal dosage of Cetuximab-IRDye800CW for fluorescence guided surgery, in comparison to the standard of care (SOC), 5-ALA fluorescent imaging agent. The main research objectives of this study are:

1. To determine the optimal dosage of Cetuximab-IRDye800CW for fluorescence guided surgery
2. To assess the safety and tolerability
3. To correlate fluorescent signals measured by in vivo multispectral imaging with Cetuximab-IRDye800CW and 5-ALA with those measured by ex vivo imaging

The study population will consist of patients, aged ≥18 years, diagnosed with high-grade glioma and scheduled for surgery.

ELIGIBILITY:
Inclusion Criteria:

* Willing to adhere to the prohibitions and restrictions specified in this protocol.
* Capable of giving signed informed consent (voluntarily), indicating that the patient understands the purpose and procedures required for the study and is willing to comply with the requirements and restrictions listed in the informed consent form and in this protocol.
* Patients aged ≥ 18 years inclusive at moment signing informed consent form.
* Established high-grade glioma (glioblastoma, grade 4 according to the WHO (World Health Organization) classification) and scheduled for surgical intervention.
* Life expectancy of > 12 weeks.
* Karnofsky performance status of at least 70%.
* No clinically significant laboratory abnormalities as determined by the investigator

  o Note: one retest of lab tests is allowed within the screening window
* Female patients should fulfil one of the following criteria:

  * At least 1 year post-menopausal (amenorrhea >12 months) at screening
  * Surgically sterile (bilateral oophorectomy, hysterectomy, or tubal ligation)
  * Women >18 years of age who are fertile, need to agree to use an adequate form of contraceptives during and till 3 months after the study. Before study enrollment, a pregnancy test in blood or urine will be performed to rule out a pregnancy. In the case of an unlikely pregnancy during the study, they accept the possible maternal/ fetal risk of participation in the study.

Exclusion Criteria:

General:

* Behavioral or cognitive impairment or psychiatric disease that in the opinion of the investigator affects the ability of the patient to understand and cooperate with the study protocol
* Deprived of freedom by an administrative or court order or in an emergency setting.
* Insufficient venous access for the study procedures.
* Close affiliation with the investigator; e.g. a close relative of the investigator, dependent person (e.g. employee or student), employee of the department of Neurosurgery of the UMCG (University Medical Center Groningen), or affiliates
* Any finding in the medical examinations or medical history giving, that in the opinion of the investigator, leads to a reasonable suspicion of a disease or condition that makes treatment with the investigational drug unadvisable, or that might affect interpretation of the results of the study or render the patient at high risk for treatment complications
* Participation in an interventional clinical study within 30 days prior to tracer administration that involved treatment with any drug (excluding vitamins and minerals) or medical device

Medical conditions

* Concomitant malignancies, including metastasized colon-, rectal-, breast carcinoma, non-small cellular lung carcinoma (NSCLC); primary epithelial ovarian-, fallopian tube-, primary peritoneal- or cervical carcinoma.
* Any abnormalities in the vital signs of the patient, as judged by the investigator, as a result of which the patient cannot participate
* eGFR (based on plasma-creatinine) outside of normal range at screening or known renal impairment (≤40 mL/min).
* Current evidence or history of bacterial, viral or fungal infections within 7 days before Cetuximab-IRDye800CW administration, as judged by the Investigator.

  o T > = 38.0°C or lab confirmed viral/bacterial/fungal infection (PCR)) or symptoms suggestive of an infection)
* Any laboratory test which is abnormal, and which is deemed by the Investigator(s) to be clinically significant
* A history of anaphylaxis, history of allergic reaction(s), known allergy to one of the drugs or excipients administered as part of this study. Mild allergies without angioedema or treatment need can be acceptable if deemed not to be of clinical significance (including but not limited to allergy to animals or mild seasonal hay fever)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2023-05-05 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Optimal dosage | 1 day
  To determine the optimal dosage of Cetuximab-IRDye800CW for fluorescence guided surgery of high-grade glioma using Near- Infrared (NIR) fluorescence imaging
To assess the safety and tolerability of intravenous tracer administration by measuring/registering the number(S)AEs and SUSARs that have occurred during the duration of the trial | 4-5 days
  The (S)AEs and SUSARS will be reported according to the CTCAE v4.0
In vivo/ex vivo correlation | 1 day
  To correlate fluorescent signals measured by in vivo multispectral imaging with Cetuximab-IRDye800CW and 5-ALA with those measured by ex vivo imaging

SECONDARY OUTCOMES:
Fluorescent signals vs pathology | 1 day
  To correlate the presence of pathologically confirmed EGFR(epidermal growth factor receptor)-gene amplification with the presence of fluorescence signals, in- and ex vivo, as measured with NIR fluorescent imaging after administering Cetuximab-IRDye800CW.
DSC biomarkers | 1 day
  Correlation between DSC (dynamic susceptibility contrast) biomarkers with pathological EGFR-gene amplification status.

CONTACTS AND LOCATIONS:
Overall Officials: Rob Groen, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- UMCG, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
upon request it can be decided whether data will/can be shared with other researchers